CLINICAL TRIAL: NCT04526041
Title: Language and Music, Speech and the Human Beatbox: Theoretical Issues for Research in General and Applied Linguistics; Monocentric Exploratory Study
Brief Title: Language and Music, Speech and the Human Beatbox: Theoretical Issues for Research in General and Applied Linguistics
Acronym: HBB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2020_0017
Record Dates: First submitted 2020-04-16; First posted 2020-08-25 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Language
Keywords: Beatbox; Human beat box; Language
MeSH Terms: conditions — Language | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Professional beatboxer singer (Other): 1 professional beatboxer singer will be asked to produced different sounds while undergoing the different procedures. Researchers wil then select the most interesting sounds to be studied.
  Interventions: Other: Nasofibroscopy; Other: Electroglottography; Other: Air flow measurement + acoustic signal recording
- Experimented beatboxer singer (Other): 10 experimented beatboxer singer will be asked to reproduced the sounds record by the first subject (professional singer) while undergoing the different procedures.
  Interventions: Other: Nasofibroscopy; Other: Electroglottography; Other: Air flow measurement + acoustic signal recording; Other: Questionnaire

INTERVENTIONS:
Other: Nasofibroscopy — Laryngeal exploration performed using a flexible fibrescope while singing.
Other: Electroglottography — Electrography of glottal movement using the EG2-PCX2 system (Glottal enterprises) while singing.
Other: Air flow measurement + acoustic signal recording — Air flow measurement and acoustic signal recording while singing using the EVA2 system (SQLab-LPL, Aix en Provence, France)
Other: Questionnaire — Questionnaire on subject singing habits, the way it use and perceive the use of his body when singing.
  Arms: Experimented beatboxer singer

SUMMARY:
Beatboxing is a form of vocal percussion primarily involving the art of mimicking drum machines, using one's mouth, lips, tongue, and voice. It may also involve vocal imitation of turntablism, and other musical instruments. To produces the different sounds, the Beatboxers use their vocal apparatus in a much wider and more complex way than its use in speech. This allows them to acquire a panel of rich and varied sounds. The Human Beatbox (HBB) is a very recent subject of study in phonetics. This study offers an exploratory study of pharyngolaryngeal articulatory behaviors using nasofibroscopy and electroglottography and an aerodynamic study in order to better understand the articulatory capacities and limits of the vocal tract.

DETAILED DESCRIPTION:
HBB is characterized by two very interesting aspects (1) the complexity of the oro-pharyngo-laryngeal joints and the articulatory precision of the beatboxers and (2) the respiratory management which allows the artists to beatbox continuously without interrupting their performance. These two points, very characteristic of this technique, allow them to best imitate diverse and varied musical tones.

The Human Beatbox is still little studied and the literature on this subject is quite limited. Percussive sounds (for example imitations of bass drums, hi-hat or snare) seem to be characterized by articulatory strategies, melodic sounds (for example wind instruments, strings) seem to be based on both articulatory and phonatory strategies, and finally, electronic sounds seem to mainly use complex phonatory strategies.

Our objectives are to better understand the articulatory capacities and limits of the vocal tract at different levels (articulation capacities, sound production mechanisms, muscular and acoustic temporal relationships, strategies of efficiency...).

It is possible to find clinical applications of the Human Beatbox in the context of congenital speech disorders (for example dyspraxia) or acquired (for example oro-pharyngo-laryngeal surgery of the partial glossectomy type).

ELIGIBILITY:
Inclusion Criteria:

* Healthy subject aged 18 or over
* Beatboxer subject (singer specializing in Beatboxing)
* Absence of language impairment
* Absence of vocal pathology
* Have signed a consent form
* Be affiliated with a Health Insurance plan.

Exclusion Criteria:

* Pregnant, parturient or lactating women
* Persons deprived of their liberty: minors or adults subject to legal protection measures or out of state to express their consent
* Subjects under guardianship or under curators

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-10-16 (Actual); Primary Completion 2021-07-27 (Actual); Study Completion 2021-07-27 (Actual)

PRIMARY OUTCOMES:
Describe and understand the production mechanisms in HBB | 1 day
  Measurement of the values of air pressure (Pa) during sound productions
Describe and understand the production mechanisms in HBB | 1 day
  Electroglottography
  iii) electroglottographic and acoustic with measurements of frequency and time acoustic parameters on acoustic analysis software.
Describe and understand the production mechanisms in HBB | 1 day
  Visualisation of larynx images

SECONDARY OUTCOMES:
Study the articulation capacities of the human vocal tract and its biomechanical limits in BeatBox singers | 1 day
  Nasofibroscopy
Study the articulation capacities of the human vocal tract and its biomechanical limits in BeatBox singers | 1 day
  Oral and nasal aeromynamics measurement.
Study the articulation capacities of the human vocal tract and its biomechanical limits in BeatBox singers | 1 day
  Analysis of acoustic signal collected during laryngeal exploration
Measure aerodynamic and muscular temporal relationships to evaluate the strategies of efficiency, performance and "economy" of the structures of the vocal tract | 1 day
  Fibroscopy images compared to accoustic signal.
Measure aerodynamic and muscular temporal relationships to evaluate the strategies of efficiency, performance and "economy" of the structures of the vocal tract | 1 day
  Aerodynamic events compared to accoustic signal.
Relate the profile of the beatboxers collected by a survey and their articulation and aerodynamic capacities evaluated during the examinations | 1 day
  Qualitative comparison between an open survey and their articulation and aerodynamic capacities (fibroscopy and accoustic signal)
Evaluate the potential contributions of the study to the fields of research in linguistics of world languages, research on acquisition and / or clinical phonetics | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Lise Crevier-Buchman, Dr, Principal Investigator — Hopital Foch
Locations (1):
- Hopital Foch, Suresnes, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No